CLINICAL TRIAL: NCT00363987
Title: A Multicenter, Randomized, Open-label, Parallel-group, Diabetic Diet-controlled Study to Evaluate the Efficacy and Safety of Compound α-Keto Acid Tablet in Combination With LPD in Delaying the Progress of Type 2 Diabetic Nephropathy
Brief Title: Controlled Study to Evaluate Efficacy and Safety of α-KA Tab With Low Protein Diet (LPD) in Delaying the Progress of Type 2 Diabetic Nephropathy (DN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Naidan Luo/medical manager, Beijing Fresenius Kabi Pharmaceutical Co
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFP503
Record Dates: First submitted 2006-08-13; First posted 2006-08-15 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-08

CONDITIONS: Diabetic Nephropathy
Keywords: nephropathy with type 2 diabetes
MeSH Terms: conditions — Diabetic Nephropathies | interventions — ketosteril; Diet, Diabetic

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ketosteril®
- 2 (Other)
  Interventions: Other: diabetic diet

INTERVENTIONS:
Drug: Ketosteril® — 1 tablet Ketosteril/5kgBW/d
  Arms: 1
Other: diabetic diet — Energy 30-35 Kcal/kg BW/d + protein 0.8 g/kg BW/d
  Arms: 2

SUMMARY:
Current expert opinion based consensus guidelines recommend usage of α-Keto analogues of essential amino acids in the diet of diabetic nephropathy patients, along with restricted protein diets. This study is designed to explore whether alpha-Keto Acid supplementation with low protein diet will retard progression of type 2 diabetic nephropathy and also to assess effects of such supplemented diets on nutritional and other parameters in this patient group.

DETAILED DESCRIPTION:
Diabetic nephropathy is the most common cause for end-stage renal disease (ESRD) in Europe and America, which is directly related to rising incidence of type 2 diabetes. In addition, life lengthening of diabetic patients and ESRD patients receiving regular therapy are also important cause. According to data in the year of 1977, 40% of newly diagnosed ESRD patients in USA were caused by diabetes. Duo to enormous number and incessant increasing incidence of type 2 diabetic patients, type 2 diabetic nephropathy patients have already accounted for considerable proportion in the diabetic nephropathy patients who need dialysis. Recently in China the incidence of type 2 diabetes shows a tendency to escalate. It is expected that the number of diabetic patients will be up to 32 million in 2010.

α-Keto Acid is a product of amino acid deamination. Because it is nonnitrogenous and can accept amino to turn into the corresponding amino acid through transaminase in the body of patient with chronic renal failure, α-Keto Acid can reduce nitrogen supply, decrease urea production, stimulate protein synthesis, suppress protein decomposition, while offering adequate essential amino acids for body. Furthermore, α-Keto Acid and branched chain amino acids do not stimulate glucagon secretion and glucagon-induced cAMP secretion in liver, has no stimulating effect on hyperfiltration, thus contribute to delaying the progress of nephropathy.

It is extensively accepted that limited intake of diet protein to reduce kidney hyperfiltration and renal glomerulus internal pressure is effective in delaying the progress of nephropathy. But at present, debate exists in clinical research papers (such as MDRDS) to the role of low protein diet in delaying the progress of nephropathy. Adding compound α-Keto Acid tablet to low protein diet for patients can prevent essential amino acid deficiency and ameliorate severity of metabolism disorder, thus prevent malnutrition. Compared with standard diabetic diet, the aim of this study is to evaluate the efficacy and safety of compound α-Keto Acid tablet in combination with low protein diet in delaying the progress of nephropathy.

This is a multicentre, randomized, open-label, parallel group, diabetic diet controlled study. 240 patients who meet Inclusion/Exclusion criteria will be randomized into test groups or control groups at the ratio of 1:1. Test group will use low protein diet in combination with compound α-Keto Acid tablet, while control group will use routine diabetic diet, efficacy and safety of test group will be compared with those of control group after 1 year treatment. The study will be performed at 12 centres to ensure that at least 200 evaluable subjects are obtained.

STUDY OBJECTIVES:

* To compare the efficacy (ameliorating proteinuria and kidney injury) of compound α-Keto Acid tablet in combination with low protein diet with that of standard diabetic diet in delaying the progress of type 2 diabetic nephropathy.
* To compare the safety of compound α-Keto Acid tablet in combination with low protein diet with that of standard diabetic diet in delaying the progress of type 2 diabetic nephropathy.

Primary Endpoint: one year of treatment with Low Protein Diet plus α-Keto Acid or Diabetic Diet; Secondary Endpoint: Death, Dialysis or renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age < 75 years, regardless of sex;
* Final diagnosis of type 2 diabetes;
* Plasma glucose is under control (fasting plasma glucose<10mmol/L, glycosylated hemoglobin<8.0%) with oral glucose-lowering agents (confine to Repaglinide, α-glycosidase inhibitors, Gliquidone) and /or insulin;
* Even through RAS blocker (ACEI/ARB) is administrated at a fixed dose (the same as the starting dose, refer to appendix 4) for more than 6 weeks, blood pressure is still ≤ 160/90 mmHg;
* Patient is without dialysis and GFR is <60ml/min/1.73m2;
* Overt proteinuria is present two times within 2 weeks (urine albumin > 300mg/d in a 24-h collection)

Exclusion Criteria:

* Diabetic ketoacidosis within the last 6 months;
* Incapable of following study requirements to control diet;
* Glomerular filtration rate < 15 ml/min/1.73m2;
* Hypercalcemia or hyperkalemia (> normal upper limit);
* Other serious disease within the last 3 months;
* With obvious symptoms or signs of liver diseases, ALT or AST > two times normal upper limit;
* Severe edema or serous cavity effusion;
* Drug abuse
* Final diagnosis of malignant tumor;
* Receiving the long-term systematic steroid hormone treatment;
* Gestation already, prepares to be pregnant in the period of the trial, lactating women;
* Participate in other product clinical trial within 30 days prior to this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
changes in urine protein and GFR | one year

SECONDARY OUTCOMES:
BMI(body mass index) | one year
Blood albumin and prealbumin | one year
Plasma High sensitivity C-reactive protein level | one year
plasma lipids | one year

CONTACTS AND LOCATIONS:
Overall Officials: Shantan Lin, Principal Investigator — Shanghai Huashan Hospital
Locations (1):
- Shanghai Huashan Hospital, Shanghai, China